CLINICAL TRIAL: NCT01588171
Title: Bemiparin Versus Enoxaparin as Thromboprophylaxis Following Vaginal and Abdominal Deliveries: A Prospective Clinical Trial
Brief Title: Comparison of 2 Low Molecular Weight Heparin as a Thromboprophylaxis Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, SHAHLA KAREEM ALALAF, Assistant Professor, Hawler Medical University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Hawler Medical University
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Venous Thromboembolic Diseases
Keywords: Deep vein thrombosis; Pulmonary embolism; Low molecular weight heparin; Enoxaparin; Bemiparin
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — bemiparin; Enoxaparin

STUDY DESIGN:
Intervention Model Description: A prospective clinical trial with sequential group allocation Women eligible for participation were assigned to the three arms of the trial: the bemiparin, enoxaparin, and control groups. Based on a schema produced by a Microsoft Excel (2007) computer program, the first woman was recruited to the non intervention group (control), the second to the bemiparin group, and the third to the enoxaparin group, with this sequence repeated throughout the trial
Masking Description: A prospective non-randomized clinical trial, no masking was applied to the 3 arms of the study
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bemiparin (Active Comparator): A new second generation Low Molecular Weight Heparin
  Interventions: Drug: Bemiparin; Drug: Enoxaparin
- Enoxaparin (Active Comparator): A well known Low Molecular Weight Heparin
  Interventions: Drug: Enoxaparin
- control group (No Intervention): Participants assigned to the Non-Interventional Arm will receive standard local hospital care as dictated by the attending physician and established clinical guidelines. Examples of standard care include, but are not limited to, patient rehydration protocols and support for ambulation or mobilization within the clinical setting. All standard safety and monitoring procedures will apply.

INTERVENTIONS:
Drug: Bemiparin — Bemiparin sodium 3,500 IU anti Xa/0.3 ml solution for injection in pre-filled syringe will be provided for each patient in Bemiparin group; subcutaneously 6 hours after delivery(vaginal and Caesarean)and then daily for up to 7 days.
  Other Names: Hibor; Laboratories Rovi Pharmaceuticals
  Arms: Bemiparin
Drug: Enoxaparin — Enoxaparin sodium 40mg (equivalent to 4,000 IU anti-Xa activity) in 0.4ml water for injection will be administered subcutaneously 6 hours after the delivery( vaginal or abdominal)then daily up to 7 days post partum, for Enoxaparin group of patients.
  Other Names: Clexane(Sanofi aventis)
  Arms: Bemiparin; Enoxaparin

SUMMARY:
The use of a new generation low molecular weight heparin (Bemiparin)and the well known LMWH (Enoxaparin) after Caesarean sections and vaginal deliveries in a risky group patients for venous thrombosis.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) is the leading cause of maternal mortality and morbidity in the developed and developing world. Pulmonary embolism and deep vein thrombosis are the two components of a single disease called deep vein thrombosis (DVT). Pregnancy associated with an average 5 to 10 fold increase in the risk of VTE compared with non-pregnant women. The highest incidence occurring during the post partum period. There are many researches done a broad on the effect of LMWH to decrease the incidence of VTE after Caesarean section using the two LMWH (Enoxaparin and Bemiparin) alone but not in one research comparing both of them alone and both together against a control group. Also according to our knowledge there are no published literature on thromboprophylaxis after vaginal delivery

ELIGIBILITY:
Inclusion Criteria:

* Presence of risk factors for venous thromboembolism
* Any parity
* Mode of delivery:vaginal, Emergency and Elective Caesarean section
* No any contraindications for Heparin

Exclusion Criteria:

* Active antenatal or postpartum vaginal bleeding.
* Placenta previa
* Thrombocytopenia
* Sever renal or liver diseases
* Uncontrolled sever hypertension
* Any patient who is already on Heparin during pregnancy

Ages: 15 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7020 (Actual)
Dates: Start 2012-05; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism | 40 days after delivery
  compare two low molecular weight heparin (Bemiparin versus Enoxaparin) after delivery with non receiver participant for development of venous thromboembolic diseases.

SECONDARY OUTCOMES:
adverse effects | after receiving the injections and till 40 days
  bruising or pain at the site of injection,Bleeding,allergic skin reactions, itching, urticaria,wound hematoma, separation, or dehiscence

CONTACTS AND LOCATIONS:
Overall Officials: Shahla K. Alalaf, Ass.Prof, Principal Investigator — Hawler Medical University; Rojan K. Jawad, High Diploma, Study Chair — Hawler Medical University; Parez R. Muhammad, High Diploma, Study Chair — Hawler Medical University; Mahabad S. Ali, High Diploma, Study Chair — Hawler ministry of Health, Directorate of Health; Namir G. Al Tawil, Professor, Study Director — Hawler Medical University
Locations (1):
- Hawler medical university, Erbil, Kurdistan Region, Iraq

REFERENCES:
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986
- [Derived] Alalaf SK, Jawad RK, Muhammad PR, Ali MS, Al Tawil NG. Bemiparin versus enoxaparin as thromboprophylaxis following vaginal and abdominal deliveries: a prospective clinical trial. BMC Pregnancy Childbirth. 2015 Mar 28;15:72. doi: 10.1186/s12884-015-0515-2. PMID 25884460